CLINICAL TRIAL: NCT07064135
Title: Impact of Prompt Medication Adjustment and Intensive Follow-up on Achieving Lipid Targets in Patients Undergoing Carotid Endarterectomy
Brief Title: Improved Medication and Care to Achieve Lipid Targets After Carotid Surgery
Acronym: IMACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barmherzige Brüder Linz (Other)
Collaborators: Johannes Kepler University of Linz (Other)
Responsible Party: Principal Investigator, Rainer Hintenberger, Senior Physician, Department of Vascular Surgery, Barmherzige Brüder Linz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMACS-2025
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Dyslipidaemias; Carotid Artery Stenoses
Keywords: LDL-C lowering; Carotid Endarterectomy; Statins; Lipid Management; Secondary Prevention
MeSH Terms: conditions — Carotid Stenosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Follow-up (Experimental): Participants in this arm receive prompt adjustment of lipid-lowering medication to achieve target LDL-C levels, combined with intensive follow-up visits and laboratory monitoring 6-8 weeks post-surgery to optimize lipid management.
  Interventions: Behavioral: Prompt Medication Adjustment and Intensive Follow-up
- Standard Care (Active Comparator): Participants in this arm receive standard postoperative care according to current guidelines, including routine follow-up and lipid management without additional early intervention or intensive monitoring.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Prompt Medication Adjustment and Intensive Follow-up — Participants receive prompt adjustment of lipid-lowering therapy perioperatively and 6-8 weeks after carotid endarterectomy to achieve guideline-recommended LDL-C targets, combined with intensive follow-up visits and laboratory monitoring. Intensive follow-up visits and laboratory monitoring of lipid parameters are performed at 6-8 weeks and again at 12-16 weeks postoperatively to optimize lipid management.
  Arms: Intensive Follow-up
Other: Standard Care — Participants receive standard postoperative care according to guidelines, including lipid management and routine follow-up without additional early intervention or intensive monitoring. Lipid parameters are assessed only once at 12-16 weeks postoperatively.
  Arms: Standard Care

SUMMARY:
The goal of this clinical trial is to find out if patients who receive extra support stay on their cholesterol-lowering therapy and therefore have lower cholesterol levels after 4 months. Extra support means regular phone calls and close monitoring before and after carotid artery surgery. The study compares this approach to usual care.

Participants will:

Be randomly assigned to either standard care or extra support for 4 months. Receive cholesterol-lowering treatment and attend follow-up visits.

DETAILED DESCRIPTION:
Cardiovascular risk factors are one of the leading causes of morbidity and mortality worldwide. Improving these often fails due to the lack of low-threshold access to specialized medical care. Especially in vascular surgery departments with multimorbid patients, optimizing the management of risk factors-particularly cholesterol-is essential.

This exploratory randomized controlled pilot study aims to investigate the effects of pharmacological optimization of cholesterol management after carotid surgery with subsequent follow-up visits. For this purpose, 50 patients who are undergoing carotid surgery due to carotid stenosis will be randomized into two groups. In Group 1, 25 patients who have not reached the lipid target at the time of surgery will be included and re-evaluated regarding their therapy after 2 months and undergo another ambulatory cholesterol check after 4 months. In Group 2, 25 patients who also have not reached the lipid target at the time of surgery will be included and, after optimization of therapy during the hospital stay, will undergo an ambulatory cholesterol check after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years
* Diagnosed carotid artery stenosis
* Planned carotid endarterectomy
* LDL cholesterol >55 mg/dL
* Willingness to participate, documented by written informed consent

Exclusion Criteria:

* Ongoing treatment with PCSK9 inhibitors
* Carotid surgery for reasons other than stenosis (e.g., traumatic injury)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving the LDL-C target of <55 mg/dL | 12-16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Clodi, Professor, MD, Study Director — Konventspital Barmherzige Brüder Linz; Juergen Falkensammer, Associate Professor, MD, Study Chair — Konventspital Barmherzige Brüder Linz
Locations (1):
- Konventhospital Barmherzige Brüder, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not yet been determined. Sharing may be considered in the future depending on ethical approval, participant consent, and data protection regulations.